CLINICAL TRIAL: NCT05149560
Title: Ticagrelor Monotherapy After Coronary Stenting in Patients With Acute Myocardial Infarction - A Prospective Single-centre, Single-arm Phase II Study
Brief Title: Ticagrelor Monotherapy After Stenting
Acronym: TIMO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number: 2021-000823-11
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Intervention Model Description: Single-centre, single-arm, prospective phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ticagrelor (Experimental): Ticagrelor 90 mg twice daily for 12 months
  Interventions: Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — All patients will be prescribed ticagrelor as monotherapy

SUMMARY:
A pilot study planned to evaluate initial safety of ticagrelor monotherapy after coronary stenting due to acute myocardial infarction.

The study is a single-centre, single-arm, prospective phase II study 200 patients who undergo coronary artery stenting due to NSTEMI or STEMI will be included.

Primary endpoint (variable):

The composite of cardiac death, spontaneous myocardial infarction or definite or probable stent thrombosis within 3 months.

DETAILED DESCRIPTION:
A pilot study with 200 subjects undergoing coronary stenting due to NSTEMI or STEMI.

All patients will undergo invasive coronary angiography and clinically indicated Percutaneous Coronary Intervention (PCI). PCI will be performed using EES and OCT guidance using the MLDMAX algorithm (Morphology, Length, Diameter, Medial dissection, Apposition, Xpansion). Eligibility criteria will be assessed after completion of PCI.

Patients will be given a drug diary to document and as a reminder of the twice daily ticagrelor administration.

The Data Safety Monitoring Board (DSMB) will continuously review the outcomes for these patients. After the first 50 patients have been recruited and at least 30 of these patients have reached 3-month follow-up or had the primary outcome, the DSMB will convene to decide whether it is safe to proceed with the study. However, the DSMB will strongly consider early termination of the trial if more than 10 primary endpoint events occur.

Patients may be treated with aspirin prior to coronary angiography, as per local treatment guidelines. All patients will be followed for 1 year. After one year, all patients will be treated per the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years old.
2. Pre- or intra-procedure treatment with ticagrelor.
3. Coronary stenting with an everolimus-eluting stent (EES) due to NSTEMI or STEMI, with post-procedure diameter stenosis <50% and post-procedure Thrombolysis In Myocardial Infarcton (TIMI) flow grade 3.
4. PCI guided by optical coherence tomography (OCT) with MLDMAX workflow
5. Subject has not yet received any post-procedure dose of aspirin or any post-procedure dose of a different P2Y12 inhibitor than ticagrelor (loading dose or pre-PCI maintenance dose of aspirin and/or a different P2Y12 inhibitor is allowed)
6. Subject has signed and dated the informed consent form.

Exclusion Criteria:

1. Planned PCI or any planned surgical intervention within the next 6 months.
2. Any indication for chronic anticoagulant therapy
3. Positive COVID-19 antigen or PCR test regardless of symptoms
4. History of definite stent thrombosis
5. Left main coronary artery stenting.
6. Stent thrombosis/restenosis as a culprit lesion.
7. Visible thrombus on angiography after PCI
8. Usage of glycoprotein IIb/IIIa inhibitors
9. Any bifurcation lesion with stenting of both branches.
10. Any treated lesion within an arterial or venous graft.
11. Any additional lesion(s) that need(s) a staged revascularization.
12. Known ejection fraction <30%.
13. Known severe renal insufficiency (eGFR <30 ml/min/1.72 m2).
14. Any life-threatening conditions or medical comorbidity resulting in life expectancy < 12 months.
15. Participation in any investigational study that has not yet reached its primary endpoint, and for which monotherapy with ticagrelor may affect the primary outcome (as per the judgement of the investigator).
16. Patients who medicate with a potent CYP3A4 inhibitor (e.g. ketoconazole, clarithromycin, nefazodone, ritonavir and atazanavir)
17. Pregnancy or woman of childbearing potential who is not sterilized or using a medically accepted form of contraception.
18. Expected inability (by the investigator) to comply with the protocol
19. Subjects incapable to giving consent personally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event | within 3 months
  The composite of cardiac death, spontaneous myocardial infarction or definite or probable stent thrombosis.

SECONDARY OUTCOMES:
Number of Participants with bleeding | within 12 months
  Bleeding Academic Research Consortium (BARC) types 3 or 5 bleeding (time-to-event)
Number of Participants with stent thrombosis or target vessel myocardial infarction | within 12 months
  Definite or probable stent thrombosis or spontaneous target vessel myocardial infarction (time-to-event)
Number of Participants with myocardial infarction | within 12 months
  Any spontaneous myocardial infarction (time-to-event)
Number of Participants that died | within 12 months
  All-cause mortality (time-to-event)
Number of Participants with major adverse cardiac event | within 12 months.
  The composite of cardiac death, spontaneous target vessel myocardial infarction or definite or probable stent thrombosis
Platelet reactivity | at 24 hours
  Platelet reactivity as assessed by the ADP-test (multiplate).
Platelet reactivity | at 3 months
  Platelet reactivity as assessed by the ADP-test (multiplate)

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Angerås, MD, PhD, Principal Investigator — Sahlgrenska Universitetssjukhus
Locations (1):
- Kardiologen, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No